CLINICAL TRIAL: NCT05074771
Title: RIabilitazione di Pazienti COvid e Loro Monitoraggio IN Casa Con la pIattaforma ARc-IntEllicare - (RICOMINCIARE)
Brief Title: At Home REhabilitation and Monitoring of People in poST-covid Condition Through ARc-inTellicare Platform (RESTART/RICOMINCIARE)
Acronym: RICOMINCIARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camlin Ltd (Industry)
Collaborators: Università Politecnica delle Marche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RICOMINCIARE
Record Dates: First submitted 2021-10-08; First posted 2021-10-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Post-COVID19; Parkinson Disease
Keywords: COVID19 Parkinson Home Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARC intellicare (Experimental): Study participants will use ARC intellicare at home, to carry out usability tests and a collection of useful data in order to optimise the system. After enrolment and training session, patients will receive an ARC unit to be used autonomously for the following 30 days.
  45 minutes 5 days / week for 4 weeks of personalized training will be carried out by the enrolled subjects: 4 weekly sessions will be unsupervised, while one will be supervised remotely by a therapist in telepresence, thanks to the integrated audio-video channel.
  Interventions: Device: ARC intellicare

INTERVENTIONS:
Device: ARC intellicare — ARC is a system that allows home motor and respiratory rehabilitation. The system includes 5 inertial measurement units for limbs and neck, a tablet with a dedicated app installed, to acquire and monitor the exercises performed by the patient in his/her daily rehab activity. Sensors and tablet can be charged on the base station. ARC allows the therapist to tailor the individual rehab project, with the support of a monitoring dashboard. The artificial intelligence engine analyses data coming from sensors positioned on the limbs, providing real-time feedback to the patient on the correct number of repetitions performed for each exercise. ARC allows therapists to create new exercises and/or select exercises from the ARC library to customize treatment (including tutorials and tips) based on condition-specific validated protocols and best practice. Patients can safely perform home rehabilitation sessions by wearing sensors and following video tutorials and tips from the ARC library.

SUMMARY:
The RESTART/RICOMINCIARE study is a pilot single-center, not controlled prospective, pre-post intervention study aimed at verifying feasibility and safety of a device-supported home rehabilitation for people suffering from mild to moderate disabilities due to respiratory or neurological conditions, related to Covid-19 or frailty condition (i.e. Parkinson Disease).

DETAILED DESCRIPTION:
The RICOMINCIARE project aims at contributing to the Covid-19 pandemic emergency by promoting the health and recovery of people recovering from Covid-19 and supporting frail people, providing an innovative telemedicine solution for the continuity of rehabilitation, able to promote and monitor remote physical rehabilitation activities in the elderly in isolation and remission from Covid-19, while containing the risk of spreading the infection. Between the people suffering from Covid-19, 80% show symptoms and 32% need hospitalization. It is estimated that the most severe cases (about 20%) have functional sequelae that persist for more than 6 months after diagnosis. In consideration of the absence of a vaccine or specific therapy, social distancing represents the main tool for limiting the infection. The use of tele-medicine is recommended and useful for everyone to ensure continuity of care in terms of monitoring, prevention and treatment

Primary objectives: to test the feasibility of integrating the ARC-Intellicare solution into the care pathway for Covid-19 survivors or frail people in terms of:

(i) adherence to the home rehabilitation program (ii) safety of rehabilitation therapy Secondary objectives: to investigate the (iiI) usability and acceptability of the intervention; (iv) the process and resources required for the new care pathway. The rehabilitation will take place according to the Good Clinical Practice (GCP) and the available guidelines regarding rehabilitation protocols and clinical and functional assessment for chronic respiratory syndromes, Post-Covid-19 conditions and neurological diseases related disabilities. Therefore, participants will undergo pre-post intervention monitoring of the clinical and functional status in terms of independence in the activities of daily life, endurance, fatigue, emotional state, quality of life following GCP.

Study design. The RICOMINCIARE study will be a pilot single-center, not controlled prospective, pre-post intervention study aimed at verifying feasibility and safety of a device supported home rehabilitation for people suffering from mild to moderate disabilities due to respiratory or neurological conditions possibly related to Covid-19.

Population. 5-10 people will be enrolled in the study between subjects who consecutively refers themselves to the study participating clinical center (Università Politecnica delle Marche, Dipartimento di Medicina Sperimentale e Clinica, Ancona) for rehabilitation management of a post-COVID-19 condition or in frailty.

A) Post-Covid-19 people: at home post-COVID-19 volunteers (discharged from hospital at home or treated at home) who have recovered from SARS-COV-2 infection (healing = two 24-hour consecutive oropharyngeal tampons negative for SARS-COV-2) from at least 15 days B) Frail people who score 9-12 on the Edmonton Frail Scale (EFS) due to neurological lesions of the motor system (i.e. Parkinson's Disease) or respiratory syndrome (COPD, pulmonary fibrosis...). Individuals should have no signs of ongoing pneumonia.

Intervention. The two-month study involves the recruitment of at least 20 patients who will use ARC-Intellicare at home, to perform usability tests and a collection of useful data in order to optimize the system.

Subsequently, the same patients will each receive an ARC-Intellicare unit for home use, to be used independently for the next 30 days.

45 minutes 5 days / week for 4 weeks of personalized training will be carried out by the enrolled subjects: 4 weekly sessions will be unsupervised, while one will be supervised remotely by a therapist in telepresence, thanks to the integrated audio-video channel.

Primary Endpoints. The primary endpoints are an adherence rate of 80% (+/- 5%) and a rate of participants' attrition (expected dropouts) of no more than 15%. The reasons for dropout or interruptions and side effects (number and types of adverse events related to the use of ARC) will also be monitored

Secondary endpoints. Secondary endpoints are a System Usability Scale (SUS) score administered to participants and informal health care workers or health care workers> 70 (i.e., the solution has a good level of usability) and a patient satisfaction of at least 80% on average on visual analog scale

Assessment timing. The entry variables and the clinical-functional data, according to the GCP, are acquired at enrolment / baseline assessment (T0) or within 7 days from the start of home intervention and at the end of the 30 days of intervention (T1), when monitoring of the primary and secondary outcome measures on adherence, acceptability and safety will be completed.

ELIGIBILITY:
Inclusion Criteria:

A) Post-Covid-19 people: at home post-COVID-19 volunteers who have recovered from SARS-COV-2 infection (healing = two 24-hour consecutive oropharyngeal tampons negative for SARS-COV-2) from at least 15 days B) Frail people who score 9-12 on the Edmonton Frail Scale (EFS) due to neurological lesions of the motor system (e.g., Parkinson's Disease) or respiratory syndrome (e.g., COPD, pulmonary fibrosis)

All subjects have to meet the following criteria:

1. Men and women> 18 years,
2. Moderate dyspnea in activities of daily living (ADL) (Barthel's dyspnea score ≤55) or walking difficulties or upper limb disabilities due to central or peripheral neurological lesions that, eventually, emerged following Covid-19 or Walking Handicap Scale (Perry and Garrett '95) ≤ 5
3. Informed consent signed

Exclusion Criteria:

1. Fever (TC ≥ 37 ° C)
2. Cough, cold, sore throat, diarrhoea or pneumonia signs and diagnosis
3. People with moderate to severe cognitive impairment (MoCA <20)
4. Formal rehabilitation performed in the last month
5. Pre-existing disability related to neurodegenerative disorders or severe stroke (TACI); epilepsy, seizures and a history of severe dizziness and falls.
6. Severe non-stabilized comorbidities: oncological diseases in the active phase; NYHA stage IV congestive heart failure; severe respiratory failure requiring cough and support for breathing; life expectancy of less than 6 months.
7. Moderate or severe dependence in activities of daily living for any medical reason (such as the participant's inability to notice or suspect to comply with the protocol procedure) or other reason the investigator believes the participant is ineligible to study (Rankin mod. ≤ 8. Women of childbearing potential who are not using suitable valid methods of contraception

9. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Adherence Rate | Daily evaluation performed on each patient using ARC during 30-day study period
  Adherence to home rehabilitation program with ARC intellicare. The adherence rate is calculated as a percentage of the number of sessions performed at home by the patient compared to the maximum number of rehabilitation sessions prescribed with ARC.
Device-related adverse events | Through study completion (8 months)
  Number and type of device-related adverse events reported
Attrition rate | Through study completion (8 months)
  % of patients who discontinue the study before the 30-day intervention period

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Pre (baseline) and post-intervention (30 days after)
  The System Usability Scale (SUS) provides a reliable tool for measuring the usability of a device. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
Patient Satisfaction | Pre (baseline) and post-intervention (30 days after)
  Visual Analogue Scale (VAS) to assess patient's satisfaction in the use of ARC
Resource consumption | Through study completion (8 months)
  Quantification of the time allocated by each healthcare professional involved in the study, from patient training on the use of ARC until the end of the study, including intermediate visits and telephonic/remote support.

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Ceravolo, Prof., Principal Investigator — Università Politecnica delle Marche, Ancona
Locations (1):
- Università Politecnica delle Marche, Ancona, Italy